CLINICAL TRIAL: NCT03513042
Title: Early Response Evaluation of Proton Therapy by PET-imaging in Squamous Cell Carcinoma Located in the Head and Neck
Acronym: ERM-PT-HNSCC
Status: Terminated | Type: Observational
Why Stopped: Inclusionrate dropped due to changes in clinical process
Sponsor: Leiden University Medical Center (Other)
Collaborators: HollandPTC (Industry)
Responsible Party: Principal Investigator, Dennis Vriens, MD, PhD, Dennis Vriens, MD, PhD (Study Coordinator), Leiden University Medical Center
Other Study IDs: NL63825.058.17; 916.18.008 (Other Grant/Funding Number: The Netherlands Organisation for Health R&D (ZonMW)); P17.291 (Other: MREC LUMC)
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: intensity-modulated proton therapy; therapy response evaluation; positron emission tomography (PET); hypoxia; metabolism; 18F-fluoroazomycin-arabinoside (FAZA); 18F-2-fluoro-2-deoxy-D-glucose (FDG); head and neck neoplasms; image-guided proton therapy; treatment outcome; predictive biomarker
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Hypoxia; Head and Neck Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Intervention:
  - Standard of care Intensity Modulated Proton Therapy (IMPT) +/- Chemotherapy.
  Baseline measurements:
  - All patients undergo baseline FDG PET-CT and FAZA PET-CT of the head-neck area.
  Interim measurements conventional):
  * FDG PET-CT will be repeated at the end of the second week of IMPT.
  * FAZA PET will only be repeated at the end of the second week of IMPT if a hypoxic tumour volume was found at baseline scanning.
  * A subcohort will also undergo activation PET imaging three times during IMPT.
  Interventions: Radiation: Intensity Modulated Proton Therapy (IMPT) +/- Chemotherapy

INTERVENTIONS:
Radiation: Intensity Modulated Proton Therapy (IMPT) +/- Chemotherapy — Standard of care:
  * IMPT (conventional fractionation [35x1,55/2Gy, 5 fractions/week] or accelerated fractionation [35x1,55/2Gy, 6 fractions/week])
  * with or without concurrent cisplatin (100 mg/m2 [d1, d22 and d43] or 40 mg/m2 weekly) or cetuximab (weekly 400 mg/m2 in 2h followed by 250 mg/m2 in 1h)

SUMMARY:
The goal of this project is to develop and characterise an imaging strategy for biology-guided individualisation of the proton therapy plan to improve patient outcome and quality-of-life.

Positron-emission tomography (PET) studies reflecting glucose metabolism, hypoxia and physical changes of proton-irradiated tumour tissues will be performed. Patients with head and neck cancer will be studied, as these individuals frequently experience recurrences within the radiation field, often with limited therapeutic options. Severe side-effects and functional impairment, deteriorating patients' quality-of-life, limited the use of dose-escalation in recent feasibility studies of photon therapy guided by individual PET-response. However, proton therapy, currently being introduced in the Netherlands, improves the precision of radiotherapy and thereby limits the side-effects caused by irradiation of neighbouring healthy tissues. Therefore, in proton therapy dose-escalation to improve patient outcome is less restricted by toxicity.

Using PET-studies of two hallmarks of radioresistance, glucose metabolism and hypoxia, side-by-side, before and early in-treatment, the predictive ability of both PET-techniques for local recurrence-free survival will be compared. A treatment plan adapted to the individual response measured by both procedures and compute tumour-dose and toxicity, will be simulated, thereby substantiating feasibility of image-guided adaptive replanning. Simultaneously to biological responses, proton therapy-induced physical changes will be studied. These atomic changes, dependent on tissue-composition and dose-deposition, are measurable by PET. It is expected that activation-PET to measure tissue-changes during therapy, a potential new biomarker of treatment efficacy, toxicity but also accuracy of treatment plan execution. Activation-PET will be related to earlier-mentioned PET-imaging of metabolism.

This clinical-technological project paves the way for an interventional trial of PET-guided treatment personalisation. Activation-PET will also serve as biomarker and quality control for proton therapy and support the current development of specialised in-beam PET-technology. These PET-techniques together will help us to individualise treatment, which is of great importance for the success and cost-effectiveness of proton therapy.

DETAILED DESCRIPTION:
Rationale: Proton therapy (PT), currently being introduced in the Netherlands, delivers radiation dose more conformal than photon radiotherapy, therefore healthy tissue damage is expected to be lower and at least similar tumouricidal effects are described. This increases the therapeutic window of radiotherapy which could be used for intensified treatment to patients prone to locoregional failure. From photon radiotherapy it is known that stratification of patients with head and neck squamous cell carcinoma (HNSCC) is possible using different positron-emission tomography (PET-)techniques. Distribution of tumour hypoxia, a main cause of resistance to radiotherapy, and glucose metabolic need have been described. PT, in contrast to photon therapy, results in activation of endogenous atoms in the irradiated tissues which can be measured using PET and reflect dose deposition and tissue composition. This provides a unique application of PET in this treatment modality as quality assurance of proton therapy and potentially as biomarker of tissue response to proton therapy. The main hypothesis is that early during PT, PET is capable of discerning a subset of patients with increased risk of locoregional failure with a univariate hazard-ratio of at least 4.0. At this time point, treatment intensification would still be possible.

Objective: To assess whether early changes in hypoxia between baseline and in the (end of the) second week of proton therapy are predictive for time-to-local recurrence in patients with HNSCC (primary). Secondary objectives include: to compare the role of hypoxia-PET to more readily available PET of glucose metabolism, to describe spatial conformity between the PET-scan and the location of the recurrence, to determine the potential of adaptive replanning based on two-timepoint PET-imaging. In a pilot setting the feasibility of activation PET in a clinical setting for quality assurance of PT-plans and potential biomarker of PT-induced tissue changes will be explored.

Study design: Prospective, single-arm, observational cohort study with invasive measurements.

Study population: Adults diagnosed with primary, unresected invasive HNSCC, planned for PT ± systemic therapy with curative intent with at least one measurable lesion larger than 2 cm at baseline (n=40).

Intervention: All patients are asked to undergo one additional baseline 18F-FAZA PET-scan (hypoxia) at baseline 18F-FDG PET-imaging (glucose metabolism) is already performed during clinical work-up. Both 18F-FAZA and 18F-FDG PET-scans will be repeated in the (end of the) second week of PT, unless no hypoxia is witnessed at baseline, then only the 18F-FDG PET-scan is repeated. In a pilot setting, 10 patients are asked to further undergo activation PET-scanning immediately after PT in the first, second and last week.

Main study parameters/endpoints: The main study parameters are the percent change in hypoxic tumour volume between baseline PET and interim PET of hypoxia and the percent change in total lesion glycolysis between baseline PET and interim PET of glucose metabolism. The primary endpoint is 3-year local recurrence-free survival (LRFS).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Each PET-acquisition will be performed in radiotherapy position preferably using fixation devices (mould mask). The procedures of PET-imaging of 18F-FAZA (hypoxia) and 18F-FDG (glucose metabolism) each involve preparation (hypoxia: none, glucose metabolism: 6h fasted), intravenous injection of a radiopharmaceutical, a waiting period in solitude (hypoxia: 2 h, glucose metabolism: 1 h), followed by PET-acquisition (hypoxia: 10-20 min, glucose metabolism: 5-10 min). Occurrence of infusion-related reactions (e.g. allergy) is highly unlikely. The radiation burden attached to each of these procedures are 6.8 mSv (hypoxia) and 2.9 mSv (glucose metabolism). The pilot substudy requires immediate transfer from PT-gantry to scanner followed by a 30-min PET-acquisition three times, resulting in an additional radiation burden of ~0.5 mSv per procedure. All other procedures are part of clinical protocol. There will be no individual benefit for enrolled subjects. Financial compensation for study-related travel expenses have been arranged. However, where possible, each study procedure will be combined with a regular visit to the PT-facility.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all following criteria:

* has reached adult age (≥ 18 years) at time of signing informed consent;
* is diagnosed with primary, cytologically/histologically proven, unresected invasive HNSCC;
* has at least one measurable lesion at baseline CT/MRI larger than 2 cm in diameter;
* is eligible for and thus candidate for PT ± systemic therapy with curative intent (for locally advanced HNSCC);
* has a life expectancy of at least 3 months;
* is expected able to undergo and willing to participate in all study and clinical procedures;
* has provided legal informed consent according to ICH/GCP and national/local regulations.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be (secondarily) excluded:

* has known presence of distant metastases;
* suffers from paranasal sinus, salivary cancer, or thyroid malignancies;
* had prior chemotherapy within the last 3 years which is considered influencing tumour biology, proposed treatment or outcome (site investigator discretion);
* had previous surgical resection for the same disease;
* had any prior radiotherapy to the head and neck region within the last 3 years which is considered influencing tumour biology, proposed treatment or outcome (site investigator discretion);
* suffers any other prior (5 years) or current malignancy (except for basal/squamous cell skin cancer, lentigo maligna, surgically cured carcinoma in situ of the cervix, in situ breast cancer or incidental finding of stage T1a-T1b prostate cancer) or serious (psychiatric) disease at study entry that could affect the treatment, evaluation or outcome of current HSCC e.g. a Karnofsky Performance Score <60 / ECOG Performance Status >2 (left to the discretion of the SI entering patient in the study);
* has uncontrolled diabetes mellitus resulting in a fasting hyperglycaemia ≥11.1 mmol.L-1 (≥200 mg.dL-1) at time of 18F-FDG PET-CT and rescheduling this investigation within the set time-window is not possible. The use of short-acting insulins within 4 h of the 18F-FDG PET scan is not allowed;
* has evidence of infection localised to the neck in the 14 days prior to 18F-FDG PET-CT;
* cannot undergo each baseline PET-CT investigations within 28 days and the start of PT;
* underwent biopsy of tumour of lymph nodes in the 14 days prior to the PET-CT scan that could interfere with imaging (left to the discretion of the PI entering patient in the study);
* is unable to tolerate lying supine for the duration of a PET-CT examination;
* is known pregnant/lactating at time of PET-CT. A negative test is not obligatory;
* specific for activation PET-CT: is scheduled to be treated in Gantry-2 (nearest to PET-CT scanner), is mobile and in case of multiple beams, only patients irradiated with a maximum angle between two beams of 90º are eligible;
* suffers from (severe) claustrophobia. Low dose benzodiazepines are allowed;
* has a history of allergic reaction or hypersensitivity attributed to compounds of similar chemical or biologic composition to 18F-FDG or 18F-FAZA (extremely unlikely);
* is known with a condition resulting in high radiation sensitivity (e.g. ataxia telangiectasia, Nijmegen Breakage Syndrome, DNA LIG4-deficiency, Fanconi anaemia [68]);
* has a known adequate renal function (creatinine clearance ≥60 mL/min/1.73m2).
* is not proficient in the Dutch or English language or has access to unbiased translators that can aid in the study procedures or clinical questionnaires;
* is unwilling or unable to provide legal informed consent (e.g. incapacitated adult), a serious (mental) condition arises, which questions persistence of informed consent, or withdraws (part) of his/her informed consent;
* in case a patient already participates in another imaging study (especially when involving additional ionising radiation such as CT-imaging), the cumulative (radiation) burden should be discussed with the PI; Participation to other than routine PT schemes (paragraph 4.4) is not an exclusion criterion per se and should be evaluated case-by-case by the coordinating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the Netherlands, 85% of patients that will be treated by PT , which includes HNSCC-patients, will be selected using a model-based approach (MBA). For every potential PT-patient an in silico comparison between a PT-plan and XRT-plan will be made to determine the amount of dose to relevant organs at risk (OARs). Using models of normal tissue complication probability (NTCP), which describe the relationship between dose and the risk of complications, the difference in NTCP ( NTCP) between PT and XRT is estimated. Cases that surpass a predefined threshold and thus are expected to significantly suffer from less toxicity from PT than XRT, will be accepted for PT and form the base population of this study.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
3-year local recurrence-free survival (LRFS) | 3 years after start of IMPT
  This is defined as the length of time (days) that the patient survives since study registration without any signs or symptoms of locoregional HNSCC assessed by structured clinical and radiological (clinical) follow-up (paragraph 8.5). If at close-out date of the study, there are no signs of locoregional recurrence, the patient will be censored to the date of the most recent follow-up examination. Distant recurrence/progression and second cancers diagnosed before locoregional recurrence and death in absence of locoregional recurrence are not considered events of interest, but will be considered as competing risk events in the analysis of this endpoint. The 2-year cumulative incidence rates will be estimated from the curves and its associated 95% confidence intervals will be calculated.

SECONDARY OUTCOMES:
3-year overall survival | 3 years after start of IMPT
  similar to LRFS but 'death from any cause' will be the event of interest
3-year disease-specific survival | 3 years after start of IMPT
  similar to LRFS but 'death from HNSCC' will be the event of interest
3-year disease-free survival | 3 years after start of IMPT
  similar to LRFS but 'any recurrence (including systemic)' will be the event of interest
tumour response per RECIST | 3 years after start of IMPT
  Response Evaluation Criteria In Solid Tumours (RECIST v1.1) tumour response during structured radiological follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Vriens, MD, PhD, Study Chair — Leiden University Medical Center (LUMC)
Locations (1):
- Holland Proton Therapy Centre (HollandPTC), Delft, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
raw data will be made publicly available as required by the funding body. A datamanagement plan including public sharing is available on request.
Time Frame: to be determined
Access Criteria: to be determined

REFERENCES:
- See also: Holland Proton Therapy Centre (HollandPTC) — http://www.hollandptc.nl